CLINICAL TRIAL: NCT02754830
Title: Single-Dose, Dose-Escalation Study With LY3303560 to Evaluate the Safety, Tolerability, and Pharmacokinetics in Healthy Subjects and Patients With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild to Moderate Alzheimer's Disease
Brief Title: A Study of LY3303560 in Healthy Participants and Participants With Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16120; I8G-MC-LMDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3303560 (Experimental): Single IV infusion 7 milligram (mg), 21 mg, 70 mg, 210 mg, 700 mg, 1400 mg, 2800 mg, and 5600 mg of LY3303560 on Day 1 in healthy participants.
  Interventions: Drug: LY3303560 - IV
- Saline Solution (Placebo Comparator): Single IV infusion of saline solution to match LY3303560 on Day 1 in healthy participants.
  Interventions: Drug: Saline Solution - IV
- LY3303560 Subcutaneous (SC) (Experimental): Single SC injection of 210 mg LY3303560 on Day 1 in healthy participants.
  Interventions: Drug: LY3303560 - SC

INTERVENTIONS:
Drug: LY3303560 - IV — Administered IV
  Arms: LY3303560
Drug: Saline Solution - IV — Administered IV
  Arms: Saline Solution
Drug: LY3303560 - SC — Administered SC
  Arms: LY3303560 Subcutaneous (SC)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the study drug, LY3303560. Side effects and laboratory results will be monitored. This study will involve single doses of LY3303560 administered intravenously (IV), meaning into a vein or subcutaneously (SC), meaning under the skin.

Screening is required within 28 days before the start of the study for healthy participants and within 70 days before the start of the study for AD participants. The study requires about 16 weeks of each participant's time including a 4 day clinical research unit (CRU) admission and 10 follow-up appointments.

This is the first time that this study drug is being given to participants. This study is for research purposes only, and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females of non-childbearing potential and who have given consent and are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* AD participants must be at least 50 years of age and have diagnostic criteria consistent with either mild cognitive impairment due to AD or mild-to moderate AD and have a positive florbetapir positron emission tomography (PET) scan

Exclusion Criteria:

* Have known allergies to LY3303560, related compounds or any components of the formulation, or history of significant atopy
* Have an increased risk of seizures
* For AD participants, evidence of macrohemorrhage or greater than 4 microhemorrhage by magnetic resonance imaging (MRI)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Parexel Early Phase Unit at Glendale, Glendale, California
  - PAREXEL-Phase 1 Baltimore Harbor Hospital Center, Baltimore, Maryland

REFERENCES:
- See also: Click here for more information about this study: A Study of LY3303560 in Healthy Participants and Participants With Alzheimer's Disease (AD) — https://trials.lilly.com/ext/trial?id=I8G-MC-LMDA

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo administered as an intravenous (IV) single dose on Day 1.
- 7 mg LY3303560: 7 milligram (mg) LY3303560 single dose administered intravenously (IV) on Day 1.
- 21 mg LY3303560: 21 mg LY3303560 single dose administered IV on Day 1.
- 70 mg LY3303560: 70 mg LY3303560 single dose administered IV on Day 1.
- 210 mg LY3303560: 210 mg LY3303560 single dose administered IV on Day 1.
- 210 mg LY3303560 Subcutaneous: 210 mg LY3303560 single dose administered subcutaneously (SC) on Day 1.
- 700 mg LY3303560: 700 mg LY3303560 single dose administered IV on Day 1.
- 1400 mg LY3303560: 1400 mg LY3303560 single dose administered IV on Day 1.
- 2800 mg LY3303560: 2800 mg LY3303560 single dose administered IV on Day 1.
- 5600 mg LY3303560: 5600 mg LY3303560 single dose administered IV on Day 1.
Period: Overall Study
Arm/Group | Placebo | 7 mg LY3303560 | 21 mg LY3303560 | 70 mg LY3303560 | 210 mg LY3303560 | 210 mg LY3303560 Subcutaneous | 700 mg LY3303560 | 1400 mg LY3303560 | 2800 mg LY3303560 | 5600 mg LY3303560
Started | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6
Completed | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Placebo: Placebo single dose administered IV.
- 7 mg LY3303560: 7 mg LY3303560 single dose administered IV.
- 21 mg LY3303560: 21 mg LY3303560 single dose administered IV.
- 70 mg LY3303560: 70 mg LY3303560 single dose administered IV.
- 210 mg LY3303560: 210 LY3303560 single dose administered IV.
- 210 mg LY3303560 SC: 210 mg LY3303560 single dose administered SC.
- 700 mg LY3303560: 700 mg LY3303560 single dose administered IV.
- 1400 mg LY3303560: 1400 mg LY3303560 single dose administered IV.
- 2800 mg LY3303560: 2800 mg LY3303560 single dose administered IV.
- 5600 mg LY3303560: 5600 mg LY3303560 single dose administered IV.
- Total: Total of all reporting groups
Arm/Group | Placebo | 7 mg LY3303560 | 21 mg LY3303560 | 70 mg LY3303560 | 210 mg LY3303560 | 210 mg LY3303560 SC | 700 mg LY3303560 | 1400 mg LY3303560 | 2800 mg LY3303560 | 5600 mg LY3303560 | Total
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.0) | 41.8 (8.7) | 48.5 (10.7) | 49.8 (11.2) | 46.3 (10.3) | 46.2 (6.7) | 46.3 (12.2) | 47.0 (13.5) | 51.7 (9.6) | 40.7 (10.4) | 46.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 2 | 3 | 2 | 1 | 3 | 1 | 2 | 3 | 22
  Male | 12 | 6 | 4 | 3 | 4 | 5 | 3 | 5 | 5 | 3 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 9
  Not Hispanic or Latino | 17 | 4 | 5 | 5 | 6 | 5 | 5 | 6 | 6 | 4 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 6 | 0 | 3 | 3 | 3 | 1 | 0 | 4 | 3 | 3 | 26
  Non-Japanese | 11 | 6 | 3 | 3 | 3 | 5 | 6 | 2 | 4 | 3 | 46
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) to be Related to Study Drug Administration
Description: Number of participants with one or more SAEs considered by the investigator to be related to study drug administration. A summary of other nonserious adverse events (AEs), and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline up to 146 days
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Groups:
- 210 mg LY3303560: 210 mg LY3303560 single dose administered IV.
Arm/Group | Placebo | 7 mg LY3303560 | 21 mg LY3303560 | 70 mg LY3303560 | 210 mg LY3303560 | 210 mg LY3303560 SC | 700 mg LY3303560 | 1400 mg LY3303560 | 2800 mg LY3303560 | 5600 mg LY3303560
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time 0 to Infinity (AUC[0-∞]) of LY3303560
Description: Serum PK: AUC. Statistical analysis was not pre-specified.
Time Frame: Day 1: Predose, 0.5, 2, 4, 12, 24, 48, 72, 96, 120, 144, 360, 528, 696, 1032, 1368, 1704, 2040 hours post-dose; additionally, for 2800 mg and 5600 mg: 2712 and 3384 hours postdose
Population: All participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per millliliter(µg*hr/mL)
Arm/Group | 7 mg LY3303560 | 21 mg LY3303560 | 70 mg LY3303560 | 210 mg LY3303560 | 210 mg LY3303560 SC | 700 mg LY3303560 | 1400 mg LY3303560 | 2800 mg LY3303560 | 5600 mg LY3303560
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6
microgram*hour per millliliter(µg*hr/mL) | 863 (15) | 2570 (8) | 11300 (16) | 27100 (15) | 16700 (17) | 98000 (34) | 219000 (28) | 325000 (25) | 788000 (21)

3. Secondary Outcome: PK: Maximum Drug Concentration (Cmax) of LY3303560
Description: Serum PK: Cmax. Statistical analysis was not pre-specified.
Time Frame: as for outcome 2
Population: All participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/millliliter (µg/mL)
Groups:
- 7 mg LY3303560 7mg: 7 mg LY3303560 single dose administered IV.
Arm/Group | 7 mg LY3303560 7mg | 21 mg LY3303560 | 70 mg LY3303560 | 210 mg LY3303560 | 210 mg LY3303560 SC | 700 mg LY3303560 | 1400 mg LY3303560 | 2800 mg LY3303560 | 5600 mg LY3303560
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6
microgram/millliliter (µg/mL) | 2.78 (12) | 7.68 (24) | 41.5 (57) | 75.0 (20) | 20.9 (18) | 331 (18) | 631 (25) | 1050 (30) | 2440 (21)

4. Secondary Outcome: Pharmacokinetics (Cerebrospinal Fluid): Area Under the Concentration Versus Time Curve (AUC) of LY3303560 in Participants With Alzheimer's' Disease (AD)
Time Frame: Day 1: Predose, 0, 2, 4, 12, 24, and 36 hours post-dose
Population: Zero participants were analyzed as no AD and Mild Cognitive Impairment (MCI) participants were enrolled.
Arm/Group | 2800 mg LY3303560 | 5600 mg LY3303560
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pharmacokinetics (Cerebrospinal Fluid): Maximum Drug Concentration (Cmax) of LY3303560 in Participants With Alzheimer's' Disease (AD)
Time Frame: Day 1: Predose, 0, 2, 4, 12, 24, and 36 hours post-dose
Population: Zero participants were analyzed as no AD and MCI participants were enrolled.
Arm/Group | 2800 mg LY3303560 | 5600 mg LY3303560
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Change From Baseline in QT/QT Corrected (QTc) Interval
Description: Mean change from baseline in QT/QTc intervals using Fridericia's formula [Fridericia's corrected QT(QTcF)] from ECG monitoring.
Time Frame: Baseline, 7 days postdose
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Groups:
- Placebo: Placebo LY3303560 single dose administered IV. .
- 70 mg LY3303560: 70 mgLY3303560 single dose administered IV.
- 5600 mg LY3303560: 5600 mg LY3303560 of 5600mg administered as an IV single dose.
Arm/Group | Placebo | 7 mg LY3303560 | 21 mg LY3303560 | 70 mg LY3303560 | 210 mg LY3303560 | 210 mg LY3303560 SC | 700 mg LY3303560 | 1400 mg LY3303560 | 2800 mg LY3303560 | 5600 mg LY3303560
Number analyzed (Participants) | 17 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6
milliseconds (msec) | 2.5 (10.7) | -0.8 (14.8) | -1.0 (8.0) | -0.9 (4.0) | -0.5 (11.8) | -1.0 (14.7) | -1.4 (14.0) | 1.7 (15.2) | 5.5 (21.3) | 0.8 (10.9)

ADVERSE EVENTS:
Time Frame: Baseline up to 146 days
Groups:
- 7 mg LY3303560: 7mg LY3303560 single dose administered IV.
- 2600 mg LY3303560: 2600 mg LY3303560 single dose administered IV.
Arm/Group | Placebo | 7 mg LY3303560 | 21 mg LY3303560 | 70 mg LY3303560 | 210 mg LY3303560 | 210 mg LY3303560 SC | 700 mg LY3303560 | 1400 mg LY3303560 | 2600 mg LY3303560 | 5600 mg LY3303560
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 6/17 | 1/6 | 1/6 | 1/6 | 2/6 | 2/6 | 3/6 | 2/6 | 1/7 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | 7 mg LY3303560 (N=6) | 21 mg LY3303560 (N=6) | 70 mg LY3303560 (N=6) | 210 mg LY3303560 (N=6) | 210 mg LY3303560 SC (N=6) | 700 mg LY3303560 (N=6) | 1400 mg LY3303560 (N=6) | 2600 mg LY3303560 (N=7) | 5600 mg LY3303560 (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Planned doses of 2800 mg and 5600 mg in AD participants were not implemented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT02754830/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT02754830/SAP_002.pdf